CLINICAL TRIAL: NCT01236417
Title: Exercise Intervention in Breast Cancer Patients With Treatment-Induced Arthralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I 169310
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer; Arthralgia
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental): Subjects will be participating in a home-based flexibility and exercise program
  Interventions: Behavioral: Exercising block

INTERVENTIONS:
Behavioral: Exercising block — Exercising for 8 weeks using an elastic band

SUMMARY:
This is a pilot study of a specifically designed exercise intervention developed for breast cancer patients with aromatase-inhibitor related joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women with a history of estrogen positive breast cancer who are receiving aromatase inhibitors for at least one month.
* Patients must complain of mild to moderate arthralgia.
* Ability to understand and sign informed consent.
* Patients meet criteria for low to moderate risk for moderate exercise based oon the ACSM guidelines.

Exclusion Criteria:

* Inability to comply with study requirements.
* Metastatic breast cancer.
* Patients with orthopedic or neuromuscular disorders that preclude participation in exercise.
* Rheumatoid arthritis.
* History of MI, angina or congestive heart failure.
* Pregnant or lactating females.
* Patients that are high risk for moderate exercise based on ACSM risk classification.
* Patients who exceed minimal physical activity recommendations from the US Surgeon General's Report: Accumulation of 30 minutes or more of moderate physical activity on most days of the week.
* Morbidly obese with BMI ≥ 40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Effects of exercise | Length of study
  To assess the effect of an exercise intervention in breast cancer patients with arthralgia secondary to adjuvant treatment with aromatase inhibitors.

SECONDARY OUTCOMES:
Feasibility of Multi-institutional study | Length of the study
  To perform a pilot to access the feasibility of a multi-institutional approach

CONTACTS AND LOCATIONS:
Overall Officials: Tracy O'Connor, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States